CLINICAL TRIAL: NCT01505530
Title: A Randomized Phase 2 Placebo-Controlled Study of LY2495655 in Patients With Advanced or Metastatic Pancreatic Cancer Receiving Chemotherapy
Brief Title: A Phase 2 Study of LY2495655 in Participants With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12552; I1Q-MC-JDDG (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — landogrozumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 300 mg LY2495655 + chemotherapy (Experimental): 300 mg LY2495655 intravenous (IV) in combination with standard of care chemotherapy (investigator's choice)
  Interventions: Drug: LY2495655; Drug: Standard of Care Chemotherapy
- 100 mg LY2495655 + chemotherapy (Experimental): 100 mg LY2495655 intravenous (IV) in combination with standard of care chemotherapy (investigator's choice)
  Interventions: Drug: LY2495655; Drug: Standard of Care Chemotherapy
- Placebo + chemotherapy (Placebo Comparator): Placebo in combination with standard of care chemotherapy (investigator's choice)
  Interventions: Drug: Placebo; Drug: Standard of Care Chemotherapy

INTERVENTIONS:
Drug: LY2495655 — Intravenous (IV) treatment every 14 days while on study. Number of Cycles: until treatment options are exhausted or unacceptable toxicity develops.
  Arms: 100 mg LY2495655 + chemotherapy; 300 mg LY2495655 + chemotherapy
Drug: Placebo — Intravenous (IV) treatment every 14 days while on study. Number of Cycles: until treatment options are exhausted or unacceptable toxicity develops.
  Arms: Placebo + chemotherapy
Drug: Standard of Care Chemotherapy — Standard of care, gemcitabine-based regimen (single-agent gemcitabine or gemcitabine plus erlotinib) or FOLFIRINOX (combination chemotherapy regimen including 5-fluorouracil, leucovorin, oxaliplatin, and irinotecan). The choice of gemcitabine-based regimen or FOLFIRINOX will be determined by the investigator (based on the standard of care used at the treating institution or as directed by local regulatory authorities).

SUMMARY:
This phase 2 study is a multicenter, randomized, double-blind, placebo-controlled trial in participants with locally advanced/inoperable or metastatic pancreatic cancer, and will investigate 2 different doses of LY2495655 in combination with standard of care chemotherapy.

ELIGIBILITY:
Inclusion:

* Unresectable or metastatic pancreas cancer; participants with previous radical surgery for pancreas cancer are eligible after progression is documented
* Participants may have received previous adjuvant treatment with gemcitabine with or without radiotherapy for pancreas cancer
* ECOG (Eastern Cooperative Oncology Group) Performance status ≤ 2
* Adequate organ function
* Have an estimated life expectancy of at least 12 weeks and in the judgment of the investigator, will be able to complete at least 2 cycles of treatment
* Ability to perform the indicated functional performance measures at baseline

Exclusion:

* Prior systemic therapy for unresectable/metastatic pancreas cancer
* Any medical or psychiatric condition, orthopedic or neuromuscular conditions that could limit participation or confound study results
* Currently taking medications that are considered both muscle building and performance enhancing (for example, androgen therapies, or anabolic steroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-12; Primary Completion 2014-10 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tyler, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenatchee, Washington
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
- Israel (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kfar Saba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
- Norway (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oslo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trondheim
- United Kingdom (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge, Cambridgeshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, England
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southampton, Hants
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Acton, London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nottingham, Nottinghamshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edinburgh, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cardiff, South Glamorgan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The reasons for discontinuation listed in the participant flow are the reasons the participant discontinued treatment and a participant was considered to have "completed" the trial if they died due to any cause while on study or completed treatment and was known to be alive at the last scheduled follow-up.
Groups:
- 300 mg LY2495655 + Chemotherapy: 300 milligram (mg) LY2495655 intravenous (IV) in combination with standard of care chemotherapy (investigator's choice).
Period: Overall Study
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Started | 41 | 43 | 41
Received At Least One Dose of Study Drug | 41 | 42 | 41
Completed One Cycle of Study Drug | 29 | 27 | 31
Completed | 0 | 0 | 0
Not Completed | 41 | 43 | 41
Not completed — Progressive Disease | 19 | 17 | 18
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 8 | 6
Not completed — Physician Decision | 6 | 2 | 5
Not completed — Sponsor Decision | 1 | 8 | 7
Not completed — Death | 7 | 6 | 5
Not completed — entry criteria not met | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy | Total
Number analyzed (Participants) | 41 | 43 | 41 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (11.3) | 67.4 (10.7) | 68.4 (9.1) | 66.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 15 | 44
  Male | 25 | 30 | 26 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 3
  Not Hispanic or Latino | 20 | 19 | 27 | 66
  Unknown or Not Reported | 21 | 21 | 14 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 5 | 9
  White | 38 | 42 | 35 | 115
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) duration was measured from the date of randomization to the date of death from any cause.
Time Frame: Baseline to Death from Any Cause (Up to 23 months)
Population: All randomized participants. Participants who were alive at data cut-off for the OS analysis or lost to follow-up were censored on the last date the participant was known to be alive. Censored participants; 300 mg LY2495655 = 9,100 mg LY2495655 =13, Placebo= 16.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 41 | 43 | 41
months | 8.02 [5.95 to 10.02] | 9.82 [5.85 to 13.54] | 10.45 [8.38 to 14.49]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from date of first dose to the first observation of disease progression or death from any cause. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST version 1.1) criteria. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: Baseline to Disease Progression or Death from Any Cause (Up to 16 months)
Population: All randomized participants.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 41 | 43 | 41
months | 4.90 [3.32 to 6.01] | 6.87 [5.36 to 7.89] | 8.21 [4.99 to 9.36]

3. Secondary Outcome: Percentage of Participants With Tumor Response Rate (RR)
Description: Response rate (RR) was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria. Complete Response (CR) was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions; Partial Response (PR) was defined as having at least a 30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD) was defined as having at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase above nadir; Stable Disease (SD) was defined as small changes that did not meet above criteria.
Time Frame: Baseline to Disease Progression (Up to 11 months)
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 41 | 43 | 41
percentage of participants | 22 | 25.6 | 26.8

4. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause. Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria. Complete Response (CR) was defined as the disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 millimeters (mm). Partial Response (PR) was defined as having at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter.
Time Frame: First CR or PR to Disease Progression (Up to 11 months)
Population: All randomized participants.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 41 | 43 | 41
months | 5.86 [3.91 to 5.98] | 8.02 [3.09 to 9.63] | 9.20 [9.03 to 10.45]

5. Secondary Outcome: Change in Lean Body Mass
Description: Change in lean body mass was assessed using dual-energy x-ray absorptiometry (DXA).
Time Frame: Baseline, Cycles 3, 5, 7, 9 and 11; Day 1
Population: All participants that received at least one dose of study drug and had evaluable post-baseline measurements.
Measure: Mean (Standard Deviation); unit: grams (g)
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 41 | 42 | 41
grams (g)
  Baseline: number analyzed (Participants) | 40 | 39 | 40
  Baseline | 43742.92 (10460.69) | 44307.12 (9853.15) | 42870.99 (8971.73)
  Cycle 3: number analyzed (Participants) | 33 | 28 | 33
  Cycle 3 | 42629.79 (10263.53) | 44250.67 (11600.33) | 42282.45 (8523.35)
  Cycle 5: number analyzed (Participants) | 24 | 25 | 27
  Cycle 5 | 43121.85 (11249.28) | 45697.82 (12035.96) | 43041.45 (7649.44)
  Cycle 7: number analyzed (Participants) | 16 | 18 | 15
  Cycle 7 | 44407.02 (11685.15) | 45486.34 (11424.00) | 45997.59 (9429.50)
  Cycle 9: number analyzed (Participants) | 10 | 14 | 12
  Cycle 9 | 46879.22 (12316.64) | 43656.49 (12335.08) | 43405.26 (7217.48)
  Cycle 11: number analyzed (Participants) | 12 | 19 | 16
  Cycle 11 | 46155.53 (9984.09) | 433316.42 (11436.93) | 45667.63 (8100.86)

6. Secondary Outcome: Change in Physical Performance Measures Using Hand Grip Strength
Description: Hand grip strength (HGS) of the non-dominant hand measured using a hand dynamometer.
Time Frame: Baseline, Cycles 2, 4, 6, 8 and 10; Day 1
Population: All participants that received at least one dose of study drug and had evaluable post-baseline measurements.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 41 | 42 | 41
kilogram (kg)
  Baseline | 28.59 (11.99) | 29.00 (11.35) | 27.46 (12.54)
  Cycle 2: number analyzed (Participants) | 24 | 27 | 28
  Cycle 2 | 25.90 (13.49) | 26.70 (12.27) | 25.26 (11.80)
  Cycle 4: number analyzed (Participants) | 18 | 18 | 21
  Cycle 4 | 25.56 (13.67) | 24.47 (10.46) | 28.02 (13.10)
  Cycle 6: number analyzed (Participants) | 12 | 19 | 15
  Cycle 6 | 26.58 (9.65) | 26.32 (14.33) | 27.43 (14.01)
  Cycle 8: number analyzed (Participants) | 8 | 9 | 9
  Cycle 8 | 27.89 (11.46) | 26.22 (14.92) | 25.44 (12.05)
  Cycle 10: number analyzed (Participants) | 8 | 13 | 11
  Cycle 10 | 25.13 (13.15) | 29.23 (14.81) | 33.27 (14.25)

7. Secondary Outcome: Change in Physical Performance Measures Using the Time Up and Go (TUG) Test
Description: Time Up and Go (TUG) is a timed walking test designed to measure gait performance and balance. It measures in seconds the time taken by an individual to stand up from a standard arm chair (approximate seat height of 46 cm [18in], arm height 65 cm [25.6 in]), walk a distance of 3 meters (118 inches, approximately 10 feet), turn, walk back to the chair, and sit down.
Time Frame: Baseline, Cycles 2, 4, 6, 8 and 10; Day 1
Population: All participants that received at least one dose of study drug and had evaluable post-baseline measurements.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 41 | 42 | 41
seconds
  Baseline | 10.70 (5.06) | 10.16 (4.53) | 10.04 (4.04)
  Cycle 2: number analyzed (Participants) | 25 | 27 | 28
  Cycle 2 | 9.19 (2.60) | 10.15 (3.93) | 10.64 (4.46)
  Cycle 4: number analyzed (Participants) | 18 | 17 | 20
  Cycle 4 | 9.33 (3.23) | 12.19 (8.96) | 9.18 (2.60)
  Cycle 6: number analyzed (Participants) | 12 | 18 | 16
  Cycle 6 | 10.14 (2.02) | 8.84 (2.94) | 9.77 (3.96)
  Cycle 8: number analyzed (Participants) | 8 | 10 | 8
  Cycle 8 | 9.28 (2.51) | 7.26 (2.13) | 9.03 (4.30)
  Cycle 10: number analyzed (Participants) | 8 | 13 | 12
  Cycle 10 | 10.56 (1.40) | 7.75 (2.38) | 9.76 (5.75)

8. Secondary Outcome: Change in Physical Performance Measures Using the 6 Minute Walk Test
Description: The 6 minute walk test measured the distance walked in 6 minutes, as quickly as possible, without running.
Time Frame: Baseline, Cycles 2, 4, 6, 8 and 10; Day 1
Population: All participants that received at least one dose of study drug and had evaluable post-baseline measurements.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 41 | 42 | 41
meter
  Baseline: number analyzed (Participants) | 41 | 40 | 39
  Baseline | 351.49 (115.18) | 382.49 (131.41) | 381.62 (94.68)
  Cycle 2: number analyzed (Participants) | 24 | 26 | 25
  Cycle 2 | 368.08 (137.65) | 361.53 (143.70) | 376.31 (107.25)
  Cycle 4: number analyzed (Participants) | 18 | 14 | 17
  Cycle 4 | 379.90 (208.66) | 323.79 (140.26) | 386.48 (126.56)
  Cycle 6: number analyzed (Participants) | 11 | 15 | 15
  Cycle 6 | 354.20 (104.74) | 416.30 (102.49) | 376.45 (132.05)
  Cycle 8: number analyzed (Participants) | 8 | 10 | 8
  Cycle 8 | 365.00 (75.71) | 347.32 (203.49) | 392.13 (113.43)
  Cycle 10: number analyzed (Participants) | 7 | 13 | 11
  Cycle 10 | 308.19 (57.23) | 372.15 (172.40) | 391.41 (143.18)

9. Secondary Outcome: Change in Physical Performance Measures Using Stair Climbing Time (StC)
Description: Stair climbing time (StC) measured the ascend and descend of a flight of 12 steps (each step 18 cm high and 28 cm deep).
Time Frame: Baseline, Cycles 3, 5, 7, 9 and 11; Day 1
Population: All participants that received at least one dose of study drug and had evaluable post-baseline measurements.
Measure: Mean (Standard Deviation); unit: joule/second
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 41 | 42 | 41
joule/second
  Baseline: number analyzed (Participants) | 25 | 22 | 21
  Baseline | 211.25 (129.57) | 206.92 (110.52) | 178.25 (65.18)
  Cycle 3: number analyzed (Participants) | 23 | 20 | 19
  Cycle 3 | 203.24 (113.76) | 203.70 (87.82) | 170.49 (76.52)
  Cycle 5: number analyzed (Participants) | 12 | 16 | 14
  Cycle 5 | 230.23 (135.31) | 211.99 (93.00) | 186.55 (95.20)
  Cycle 7: number analyzed (Participants) | 11 | 9 | 9
  Cycle 7 | 198.24 (83.19) | 235.82 (111.95) | 200.79 (130.74)
  Cycle 9: number analyzed (Participants) | 5 | 8 | 5
  Cycle 9 | 217.82 (131.34) | 197.49 (102.51) | 160.59 (87.60)
  Cycle 11: number analyzed (Participants) | 6 | 6 | 1
  Cycle 11 | 193.24 (96.70) | 221.59 (107.49) | 188.78 (188.78)

10. Secondary Outcome: Change in Patient Reported Outcomes (PRO)
Description: Data from PRO scales are not be presented. An error in coding the scales (coded differently early and late in the study) occurred. Unable to determine which results were affected therefore analysis not completed.
Time Frame: Baseline, Cycles 2, 4, 6, 8 and 10; Day 1
Population: Zero participants analyzed. An error in coding the scales (coded differently early and late in the study) occurred. Unable to determine which results were affected therefore analysis not completed.
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change in Pain Scale Physical Functioning
Description: The 36-item Short-Form Health Survey (SF-36) pain scale is a generic, health-related scale assessing participant's quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). The PCS physical functioning domain score ranges from 0 to 100 (higher scores indicate better health status).
Time Frame: Baseline, Cycles 2, 4, 6, 8 and 10; Day 1
Population: All randomized participants with evaluable SF-36 domain scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 41 | 43 | 41
units on a scale
  Baseline: number analyzed (Participants) | 37 | 37 | 37
  Baseline | 6.62 (2.23) | 6.81 (2.55) | 5.89 (2.54)
  Cycle 2: number analyzed (Participants) | 21 | 24 | 26
  Cycle 2 | 4.48 (2.09) | 5.63 (2.81) | 5.04 (2.03)
  Cycle 4: number analyzed (Participants) | 18 | 18 | 18
  Cycle 4 | 5.33 (1.91) | 4.78 (2.02) | 4.83 (2.50)
  Cycle 6: number analyzed (Participants) | 8 | 17 | 16
  Cycle 6 | 4.38 (1.51) | 4.65 (2.29) | 4.25 (1.91)
  Cycle 8: number analyzed (Participants) | 7 | 13 | 10
  Cycle 8 | 4.14 (1.46) | 5.85 (2.44) | 5.00 (2.26)
  Cycle 10: number analyzed (Participants) | 7 | 12 | 11
  Cycle 10 | 4.57 (2.57) | 5.58 (2.87) | 3.55 (1.92)

12. Secondary Outcome: Number of Participants With Anti-LY2495655 Antibodies
Time Frame: Cycle 1, Day 1 and Day 29 (Pre-Dose); Cycle 6 Day 1
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg LY2495655 + Chemotherapy | 100 mg LY2495655 + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 41 | 43 | 41
Participants | 0 | 1 | 1

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug.
Groups:
- 300 mg LY2495655: 300 mg LY2495655 intravenous (IV) in combination with standard of care chemotherapy (investigator's choice).
  LY2495655: Intravenous (IV) treatment every 14 days while on study.
- 100 mg LY2495655: 100 mg LY2495655 intravenous (IV) in combination with standard of care chemotherapy (investigator's choice).
  LY2495655: Intravenous (IV) treatment every 14 days while on study.
- Placebo: Placebo in combination with standard of care chemotherapy (investigator's choice).
  Placebo: Intravenous (IV) treatment every 14 days while on study.
Arm/Group | 300 mg LY2495655 | 100 mg LY2495655 | Placebo
Serious Adverse Events (participants affected / at risk) | 26/41 | 30/42 | 25/41
Other Adverse Events (participants affected / at risk) | 41/41 | 41/42 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 300 mg LY2495655 (N=41) | 100 mg LY2495655 (N=42) | Placebo (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (8) | 4 (7) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 4 (7) | 1 (1)
Device occlusion (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (3) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (2)
Pain (General disorders) | 1 (3) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (8) | 7 (7) | 5 (8)
Bile duct obstruction (Hepatobiliary disorders) | 2 (3) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 3 (15) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (7) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (6) | 1 (3) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (10) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (5) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/16 (0) | 1/13 (5) | 0/15 (0) — This event is gender specific, only occurring in female participants. The number of participants exposed has been adjusted accordingly.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 2 (7) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 300 mg LY2495655 (N=41) | 100 mg LY2495655 (N=42) | Placebo (N=41)
Anaemia (Blood and lymphatic system disorders) | 12 (58) | 14 (63) | 19 (58)
Neutropenia (Blood and lymphatic system disorders) | 12 (35) | 9 (50) | 13 (58)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (28) | 11 (37) | 14 (46)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (10) | 3 (13)
Abdominal pain (Gastrointestinal disorders) | 12 (38) | 6 (25) | 10 (49)
Ascites (Gastrointestinal disorders) | 4 (8) | 4 (12) | 7 (22)
Constipation (Gastrointestinal disorders) | 12 (40) | 14 (57) | 9 (49)
Diarrhoea (Gastrointestinal disorders) | 22 (51) | 17 (65) | 20 (61)
Dry mouth (Gastrointestinal disorders) | 6 (20) | 4 (22) | 6 (16)
Dyspepsia (Gastrointestinal disorders) | 3 (15) | 3 (5) | 4 (14)
Flatulence (Gastrointestinal disorders) | 3 (20) | 2 (12) | 4 (12)
Mouth ulceration (Gastrointestinal disorders) | 4 (12) | 2 (10) | 2 (2)
Nausea (Gastrointestinal disorders) | 18 (54) | 19 (107) | 18 (63)
Stomatitis (Gastrointestinal disorders) | 5 (20) | 4 (9) | 4 (11)
Vomiting (Gastrointestinal disorders) | 13 (24) | 14 (32) | 14 (33)
Asthenia (General disorders) | 2 (10) | 2 (5) | 4 (13)
Chest pain (General disorders) | 3 (18) | 2 (13) | 1 (3)
Fatigue (General disorders) | 25 (131) | 28 (138) | 28 (151)
Influenza like illness (General disorders) | 5 (16) | 4 (5) | 4 (6)
Mucosal inflammation (General disorders) | 7 (26) | 6 (11) | 4 (14)
Oedema peripheral (General disorders) | 9 (46) | 14 (40) | 14 (50)
Pain (General disorders) | 5 (10) | 5 (27) | 3 (7)
Peripheral swelling (General disorders) | 4 (16) | 3 (6) | 2 (7)
Pyrexia (General disorders) | 13 (24) | 11 (41) | 13 (24)
Hypersensitivity (Immune system disorders) | 3 (4) | 1 (2) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (5)
Oral candidiasis (Infections and infestations) | 2 (2) | 1 (2) | 4 (10)
Tooth infection (Infections and infestations) | 0 (0) | 3 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 6 (10) | 4 (8)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (18) | 3 (13)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (18) | 4 (15)
Blood alkaline phosphatase increased (Investigations) | 1 (8) | 3 (16) | 3 (14)
Blood bilirubin increased (Investigations) | 3 (6) | 4 (7) | 3 (6)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (14)
Neutrophil count decreased (Investigations) | 4 (14) | 3 (4) | 5 (12)
Platelet count decreased (Investigations) | 8 (14) | 5 (15) | 4 (11)
Weight decreased (Investigations) | 9 (25) | 6 (17) | 8 (45)
White blood cell count decreased (Investigations) | 2 (2) | 3 (16) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 18 (60) | 17 (75) | 21 (103)
Dehydration (Metabolism and nutrition disorders) | 5 (7) | 3 (5) | 6 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (15) | 1 (3) | 3 (23)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (8) | 3 (5) | 5 (13)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (11) | 3 (9) | 8 (19)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (15) | 5 (13) | 2 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (18) | 3 (11) | 2 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (25) | 8 (35) | 4 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (12) | 2 (9) | 2 (12)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (23) | 1 (2) | 2 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (2) | 3 (16)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (24) | 1 (2) | 3 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (10) | 3 (18) | 5 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (26) | 1 (1) | 3 (15)
Dizziness (Nervous system disorders) | 6 (27) | 8 (36) | 4 (21)
Dysgeusia (Nervous system disorders) | 6 (23) | 5 (14) | 9 (47)
Headache (Nervous system disorders) | 6 (22) | 3 (15) | 2 (3)
Neuropathy peripheral (Nervous system disorders) | 4 (29) | 2 (15) | 5 (19)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (17) | 2 (20) | 5 (41)
Anxiety (Psychiatric disorders) | 4 (12) | 4 (28) | 2 (12)
Confusional state (Psychiatric disorders) | 4 (6) | 1 (3) | 1 (1)
Depression (Psychiatric disorders) | 4 (9) | 5 (33) | 4 (21)
Insomnia (Psychiatric disorders) | 6 (38) | 4 (20) | 1 (7)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/16 (0) | 0/13 (0) | 1/15 (1) — This event is gender specific, only occurring in female participants. The number of participants exposed has been adjusted accordingly.
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (26) | 7 (19) | 6 (21)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (14) | 1 (1) | 4 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (38) | 10 (43) | 7 (33)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (15) | 2 (5) | 4 (11)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (8) | 3 (10) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (8) | 1 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (19) | 2 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (23) | 6 (42) | 3 (35)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (6) | 2 (3) | 3 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (17) | 4 (34) | 4 (24)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (13) | 3 (11) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 6 (18) | 6 (13) | 6 (24)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (4) | 2 (2) | 4 (12)
Deep vein thrombosis (Vascular disorders) | 2 (5) | 2 (15) | 4 (8)
Hot flush (Vascular disorders) | 3 (14) | 2 (6) | 1 (5)
Hypertension (Vascular disorders) | 1 (1) | 4 (22) | 3 (8)
Hypotension (Vascular disorders) | 4 (13) | 5 (9) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days